CLINICAL TRIAL: NCT03595683
Title: Phase II Dual-Cohort Study Evaluating the Effects of Pembrolizumab in the Presence of Gut Microbiota Modulation With EDP1503 in Advanced Melanoma Naïve or Refractory to Anti-PD1 Antibody
Brief Title: Pembrolizumab and EDP1503 in Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply no longer available.
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0461
Record Dates: First submitted 2018-06-19; First posted 2018-07-23 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Melanoma (Skin); Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Anti-PD1 naive (Experimental): Participants that have not received prior anti-PD1 therapy for their cancer will be enrolled to this arm.
  Interventions: Drug: Pembrolizumab; Biological: EDP1503
- Cohort 2: Anti-PD1 refractory (Experimental): Participants that have received prior anti-PD1 therapy for their cancer will be enrolled to this arm.
  Interventions: Drug: Pembrolizumab; Biological: EDP1503

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg given by intravenous (IV) infusion once every 3 weeks.
  Other Names: Keytruda
Biological: EDP1503 — Taken by mouth twice daily. Each capsule will contain ≥ 7.5x10^10 colony-forming units (CFU).

SUMMARY:
This study is being done to determine if orally administered EDP1503 will enhance the response to standard immunotherapy treatment (pembrolizumab) in participants with advanced melanoma.

The study will involve initial administration of EDP1503 for a run-in period (2 weeks) followed by administration of both EDP1503 (twice daily) and pembrolizumab (every 3 weeks).

Mandatory biopsies are required before starting study treatment and after 2 weeks of EDP1503 dosing.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, unresectable or metastatic melanoma
* Be willing and able to provide written informed consent/assent for the trial.
* Aged 18 years or older on day of signing informed consent.
* Have measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* Be naïve to exposure in the metastatic setting to PD1/L1 antibody for cohort 1 but have had exposure to PD1/L1 (or PD1/L1 combination therapy) in cohort 2. Prior exposure to CTLA4 antibody in the metastatic setting is not allowed for cohort 1 though exposure in the adjuvant setting is allowed for either cohort. To be eligible for cohort 2, and considered refractory to PD1/L1, a patient must have had a restaging exam showing progressive disease at least 90 days following initiation of anti-PD1/L1 as prior therapy.

  * Adjuvant therapy with BRAF-MEK, PD1 or CTLA4 based therapy is allowed. Prior adjuvant BRAF-MEK therapy will fulfill treatment requirement in the metastatic setting. Patients who experience progression of disease during adjuvant PD1 therapy or within 6 months of completing adjuvant PD1 therapy will be considered refractory and thus eligible for cohort 1. Patients with progression to active metastatic disease more than 6 months following completion of adjuvant PD1 therapy will be eligible for cohort 1.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of study initiation.
* Adequate Organ Function Laboratory Values

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin >2.5 mg/dL
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. [Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.]
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. [Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.]

Exclusion Criteria:

* For cohort 2: Has BRAF mutant disease but has not yet received treatment with RAF/MEK inhibitors. This criteria can be met via adjuvant treatment with BRAF-MEK inhibitors
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks of the first dose.
* Is currently taking Bifidobacterium based probiotics or is taking pre/pro-biotics regularly.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose.
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1 (excluding anti-PD1 antibodies such as pembrolizumab or nivolumab in cohort 2) or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to start of study. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring antibiotic therapy or has received a course of antibiotics within the previous 2 weeks of starting study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days of planned start of study therapy. [Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Luke, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2018 and 2020 a total of 10 patients signed study consent from two sites. Two patients failed screening and the remaining 8 enrolled and underwent study treatment. Study was closed early due to EDP1503 no longer being manufactured.
Period: Overall Study
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Started | 3 | 5
Run-in Phase | 3 | 5
Combination Phase | 0 | 1
Completed (Treatment completed per protocol) | 0 | 1
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Pursue alternative therapy | 1 | 1
Not completed — Progressive disease | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Median (Full Range); unit: years] | 70 [63 to 74] | 59 [40 to 82] | 63 [40 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: For Cohort 1, based on deep response (>80% tumor reduction). Assessed by standard RECIST criteria for Cohort 2 (complete + partial response).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

2. Primary Outcome: Number of Participants With EPD1503 Related Adverse Events During the Run in Period
Description: Assessed by CTCAE v4.0, grade 3 or higher
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from first dose of either drug until disease progression or death from any cause. Surviving subjects without progression will be censored as of the date of the last negative examination. Estimated using the Kaplan-Meier method
Time Frame: 2 years
Measure: Median (Standard Error); unit: months
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 3 | 5
months | 8.6 (0.5) | 2.7 (0.7)

4. Secondary Outcome: Number of Participants With Treatment Related Adverse Events During Combination Therapy
Description: Assessed by CTCAE v4.0, grade 3 or higher
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 3 | 5
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: All serious adverse events are reported and other adverse events related to treatment were collected and reported here.
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Anti-PD1 Naive (N=3) | Cohort 2: Anti-PD1 Refractory (N=5)
Sepsis (Infections and infestations) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Fatigue (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Anti-PD1 Naive (N=3) | Cohort 2: Anti-PD1 Refractory (N=5)
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Fatigue (General disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Serum amylase increased (Investigations) | 1 | 0
Elevated TSH (Investigations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT03595683/Prot_SAP_000.pdf